CLINICAL TRIAL: NCT06943729
Title: Clinical Safety and Efficacy of Flow Diverter in the Treatment of Intracranial Aneurysms
Brief Title: Clinical Safety and Efficacy of Flow-diverter in the Treatment of Intracranial Aneurysms
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); Ningbo No.2 Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Second Affiliated Hospital of Nanchang University (Other); Jiangxi Provincial People's Hopital (Other); Zhengzhou Central Hospital (Other); Xuchang Central Hospital (Unknown); Second People's Hospital of Hunan (Other); People's Hospital Of Ningxiang City (Unknown); The First People's Hospital of Changde City (Other); HUANG GANG Central Hospital (Unknown); Xianning Central Hospital (Other); Jingzhou Central Hospital (Other); Yichang Central People's Hospital (Other); The First People's Hospital of Changzhou (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Northern Jiangsu People's Hospital (Other); Suzhou Municipal Hospital (Other); Jiangsu Taizhou People's Hospital (Other); Huadong Hospital (Other); RenJi Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai Fourth People's Hospital (Unknown); Shanghai Donglei Brain Hospital (Unknown); Shanghai Pudong New Area People's Hospital (Other); Shanghai East Hospital of Tongji University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Tangshan Gongren Hospital (Other); The Second Hospital of Hebei Medical University (Other); Hebei General Hospital (Other); Xingtai People's Hospital (Other); Peking University First Hospital (Other); THE AFFILIATED SUZHOU HOSPITAL OF NANJING UNIVERSITY MEDICAL SCHOOL (Unknown); The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yuxiang Gu, Vice-president of Huashan Hospital west campus, Huashan Hospital
Other Study IDs: KY2025-698
Record Dates: First submitted 2025-04-14; First posted 2025-04-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Flow Diverter
Keywords: Flow Diverter; Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To collect the safety and effectiveness data of flow-di in the treatment of intracranial aneurysms in real-world clinical practice, verify its classification of treatment strategies for aneurysms of different locations and shapes, and optimize postoperative medication regimen, provide long-term evidence-based basis for clinical treatment of intracranial aneurysms, and build a database.

DETAILED DESCRIPTION:
The purpose of this study is to verify the clinical safety and effectiveness of Flow Diverters (FD) in the treatment of intracranial aneurysms. In recent years, FD, as a new type of minimally invasive interventional treatment method, has been widely used in the treatment of various types of intracranial aneurysms. FD promotes the formation of thrombosis in the aneurysm by changing the hemodynamics of the aneurysm, and promotes the repair of vascular endothelium, thereby achieving tumor occlusion. In this study, 523 patients with various types of intracranial aneurysms will be recruited in 36 centers, using a multicenter, prospective, single-arm study design. The main goal of the study was to assess the complete occlusion rate of aneurysms in the 12 months after FD treatment. Secondary goals included postoperative complications (such as cerebral infarction, intracranial thrombosis), postoperative nerve function recovery, and patients' quality of life. At the same time, a large-scale domestic FD database for the treatment of intracranial aneurysms was established. The results of the study will verify the efficacy and safety of FD through clinical imaging evaluation (mainly cerebral angiography) and long-term clinical follow-up data. At the same time, the success rate of surgery and the incidence of restenosis in the stent are analyzed to comprehensively evaluate the application prospects of FD in the treatment of intracranial aneurysms. The results of this study will provide an important evidence-based basis for further promoting the clinical application of FD, optimizing the treatment plan of aneurysms, and improving the patient's prognosis.

ELIGIBILITY:
Inclusion Criteria:

1)18 years ≤80 years; 2) intracranial aneurysm diagnosed by CTA, MRA or DSA (Including wide-necked aneurysms (neck width ≥4mm or Dome/neck ratio <2), saccular, fusiform aneurysms, recurrent saccular aneurysms and dissecting aneurysms, and the diameter of the parent vessel ≥ 2.0 mm and ≤ 6.0 mm; the location includes: anterior circulation C3 segment and above of internal carotid artery, distal artery of Willis circle, posterior circulation V4 segment of vertebral artery and basilar artery and its main branches; 3) Voluntary participation in this study and signing of the Informed Consent Form (ICF).

Exclusion Criteria:

1)AVM related aneurysm; 2) Acute ruptured aneurysm; 3) Severe stenosis or tortuosity of intracranial artery, or anatomical abnormality, which makes it difficult for the device to reach the lesion ; 4) Patients with hemorrhagic or ischemic stroke within 30 days; 5) Modified Rankin Score (mRS)>2 points before operation; 6) Patients with life expectancy less than 12 months; 7) Patients with definite history of allergy to cobalt-chromium alloy and platinum-tungsten alloy materials; Allergy to contrast media; 8) antiplatelet (PLT)<100×10^ 9 /L or/and anticoagulation contraindicated; 9) pregnant or lactating women; 10) other study participants who were assessed by the investigator as unsuitable for participation in the study.

Intraoperative exclusion criteria: 1) acute rupture and hemorrhage of aneurysm during operation; 2) failure of FD implantation; 3) thrombosis in stent; 4) stent mal-apposition.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intracranial aneurysm diagnosed by CTA, MRA or DSA (Including wide-necked aneurysms (neck width ≥4mm or Dome/neck ratio <2), saccular, fusiform aneurysms, recurrent saccular aneurysms and dissecting aneurysms, and the diameter of the parent vessel ≥ 2.0 mm and ≤ 6.0 mm
Sampling Method: Probability Sample
Enrollment: 523 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Aneurysm complete occlusion rate 12 months after surgery | 12 months after surgery

SECONDARY OUTCOMES:
Aneurysm complete occlusion rate 6 months after surgery | 6 months after surgery
Immediate success rate | Immediate
In-stent stenosis (>50% stenosis) rate 6,12 months after surgery | 6,12 months after surgery
Incidence of ipsilateral disabled stroke 3 months after surgery, 6 months after surgery, and 12 months after surgery | 3 months after surgery, 6 months after surgery, and 12 months after surgery
neurogenic death rate 6 months and 12 months after surgery | 6 months and 12 months after surgery
Target aneurysm recurrence retreatment rate 6 months and 12 months after surgery | 6 months and 12 months after surgery
Proportion of study participants with mRS score 0-2 | 3 months after surgery, 6 months after surgery, and 12 months after surgery
Incidence of adverse events (AE) and severe adverse events (SAE) | 3 months after surgery, 6 months after surgery, and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gu Yuxiang, PhD, Study Chair — department of Neurosurgery, Huashan Hospital,Fudan University
Locations (1):
- Huashan hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No